CLINICAL TRIAL: NCT01737840
Title: Intravenous Pantoprazole vs Ranitidine in Dyspepsia in Emergency Department: A Randomized Controlled Trial.
Brief Title: Comparison of Pantoprazole and Ranitidine in Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 160
Record Dates: First submitted 2012-11-24; First posted 2012-11-30 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Dyspepsia
Keywords: dyspepsia; pantoprazole; ranitidine; emergency department
MeSH Terms: conditions — Dyspepsia; Emergencies | interventions — Pantoprazole; Ranitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pantoprazole (Experimental): Intravenous pantoprazole 40 mg flacon
  Interventions: Drug: Pantoprazole
- ranitidine (Active Comparator): Intravenous ranitidine 50 mg
  Interventions: Drug: Ranitidine

INTERVENTIONS:
Drug: Pantoprazole — 33 patients
  Other Names: Pantpas
  Arms: pantoprazole
Drug: Ranitidine — 33 patients
  Other Names: Ulcuran
  Arms: ranitidine

SUMMARY:
The H0 hypothesis of the study is there is no difference between pantoprazole and ranitidine in treating patients presented with dyspepsia to the emergency department.

The H1 hypothesis is there is difference between pantoprazole and ranitidine in treating patients presented with dyspepsia to the emergency department.

DETAILED DESCRIPTION:
Dyspepsia is one of the common complaints in emergency department. Proton pomp inhibitors, H2 receptor blockers and anti-acids are common drugs for treating dyspepsia in emergency department. However there is no study in the emergency department comparing the effectiveness of these drugs. So the investigators planned this study which drug is effective in these patients in order to provide a cost-effective treatment in dyspeptic patients.

ELIGIBILITY:
Inclusion Criteria:

* Epigastric pain
* Older than 18 years old

Exclusion Criteria:

* Diagnosed as cholecystitis, pancreatitis, myocardial infarction, etc.. at the end of the emergency deparment evaluation period.
* Pregnancy
* Patients with unstable vital signs
* Patients used anti-acid, H2 receptor blockers and proton pomp inhibitors in the last one hour.
* Allergy to H2 receptor blockers and proton pomp inhibitors.
* Patients denied to give inform consent and who are illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cenker Eken, Proffesor, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Welling LR, Watson WA. The emergency department treatment of dyspepsia with antacids and oral lidocaine. Ann Emerg Med. 1990 Jul;19(7):785-8. doi: 10.1016/s0196-0644(05)81704-4. PMID 2202240
- See also: The web adress of the organization which this study is conducted. — http://www.akdeniz.edu.tr

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pantoprazole | Ranitidine
Started | 35 | 35
Completed | 33 | 33
Not Completed | 2 | 2
Not completed — Diagnosed with an other pathology | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole | Ranitidine | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 66
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (16.4) | 34.8 (13.9) | 36.6 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 15 | 11 | 26
Region of Enrollment [Number; unit: participants]
  Turkey | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale Score
Description: The investigators are measuring the change of pain from the baseline to the 30th and 60th minutes by visual anologue scale (VAS). Visual Analogue Scale measurement is between 0 (no pain) and 100 (worst pain). A decrease of 13 or 16 mm in VAS score is accepted as a minimum clinically significant change in pain.
Time Frame: 30th and 60th minutes
Measure: Mean (Standard Deviation); unit: Visual Analogue Scale
Groups:
- Pantoprazole: Intravenous pantoprazole 40 mg
Arm/Group | Pantoprazole | Ranitidine
Number analyzed (Participants) | 33 | 33
Visual Analogue Scale
  VAS score changes at 60 minutes | 39.6 (39) | 42.3 (25)
  VAS scores changes at 30 minutes | 27.6 (28) | 28.3 (23)

2. Secondary Outcome: Need for Additional Drug
Description: The investigators are measuring the need for additional drug at the end of 60 minutes.
Time Frame: 60 th minute
Measure: Number; unit: participants
Arm/Group | Pantoprazole | Ranitidine
Number analyzed (Participants) | 33 | 33
participants | 13 | 8

ADVERSE EVENTS:
Time Frame: 60 minutes
Arm/Group | Pantoprazole | Ranitidine
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No